CLINICAL TRIAL: NCT01485562
Title: Treatment of Postpartum Haemorrhage (PPH) Using Misoprostol in Home Births
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Aga Khan Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.4.15
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Haemorrhage
Keywords: postpartum haemorrhage; misoprostol; treatment; prophylaxis; home births
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): women who experience a PPH will be randomized to receive 800 misoprostol (four tablets of 200 mcg administered sublingually)
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): women who experience a PPH will be randomized to receive 4 placebo tablets administered sublingually
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Misoprostol — 4 tablets of 200 mcg misoprostol administered sublingually if the woman experiences a PPH after child birth
  Other Names: Gymiso
  Arms: Misoprostol
Other: placebo — 4 tablets, administered sublingually if the woman experiences a PPH
  Other Names: Gymiso
  Arms: placebo

SUMMARY:
A double-blind individual randomized controlled study of misoprostol vs. placebo for treatment in homebirths in the Chitral district, in the Khyber Pakhtunkhwa province in Pakistan.

DETAILED DESCRIPTION:
A double-blind individual randomized controlled study of misoprostol vs. placebo for treatment in homebirths in the Chitral district, in the Khyber Pakhtunkhwa province in Pakistan. The purpose of the study is to assess the overall clinical and programmatic effectiveness of Traditional Birth Attendants (TBAs) administering 800 mcg sublingual misoprostol to treat Postpartum Haemorrhage (PPH) at the community level.

The study will recruit pregnant women who deliver at home. All women enrolled in the study will receive misoprostol for prevention (600 mcg oral dose). Women diagnosed with PPH will be randomized to receive either a) standard care + 800 mcg sublingual misoprostol (four 200 mcg tablets) or b) standard care + four placebo tablets resembling misoprostol. In this setting, standard care is uterine massage and/or compression and referral to the nearest health facility or attendance by the Lady Health Visitor/ Community Health Nurse.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver at home with a study TBA present.
* Women must be willing and able to provide informed consent
* Women must agree to participate in a follow up interview
* Women must agree to have pre and post-partum haemoglobin taken

Exclusion Criteria:

* If the woman does not meet any of the above outlined inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Haemoglobin concentration (Hb) of greater than or equal to 2 g/dl from pre- to post-delivery | 3-5 days after delivery
  The primary outcome will measure the proportion of women who experience a drop in their haemoglobin concentration (Hb) of greater than 2 g/dl from pre- to post-delivery.

SECONDARY OUTCOMES:
Number of participants who experience side effects | immediately after delivery; 3-5 days post delivery
  number of women who experienced side effects and the severity of the side effects as rated on a scale, additional care provided
number of participants who received additional interventions | immediately after delivery; 3-5 days post delivery
  number of participants who received care by as skilled provider and the type of care provided
number of women who found misoprostol treatment to be acceptable | immediately after delivery; 3-5 days post delivery
  women will be asked to rate their acceptability with the treatment using a scale
number of participants who experience severe adverse events | immediately after delivery; 3-5 days post delivery
  serious adverse are defined as uterine rupture, hysterectomy, hospitalization, maternal deaths, and neonatal deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Zafar Khan, Principal Investigator — Aga Khan Health Services; Nadeem Zuberi, Study Director — Aga Khan University; Gijs Walraven, Study Director — Secretariat of His Highness the Aga Khan, Aiglemont; Ayisha Diop, Study Director — Gynuity Health Projects; Dina Abbas, Study Director — Gynuity Health Projects
Locations (1):
- Home Births, Chitral, Khyber Pakhtunkhwa, Pakistan

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518
- [Derived] Abbas DF, Jehan N, Diop A, Durocher J, Byrne ME, Zuberi N, Ahmed Z, Walraven G, Winikoff B. Using misoprostol to treat postpartum hemorrhage in home deliveries attended by traditional birth attendants. Int J Gynaecol Obstet. 2019 Mar;144(3):290-296. doi: 10.1002/ijgo.12756. Epub 2019 Jan 24. PMID 30582753